CLINICAL TRIAL: NCT05724251
Title: Effect of Iodine Deficiency on Periodontitis
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Didem OZKAL EMINOGLU, assistant professor, Ataturk University
Other Study IDs: 9375
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Periodontal Diseases; Periodontitis; Iodine Deficiency; Periodontitis, Adult
Keywords: periodontitis; Iodine Deficiency
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — urine of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: participants without periodontitis
  Interventions: Other: healthy
- periodontitis: participants with stage-3 periodontitis
  Interventions: Other: periodontitis

INTERVENTIONS:
Other: healthy — no intervention
  Groups: Healthy
Other: periodontitis — no intervention
  Groups: periodontitis

SUMMARY:
The goal of this observational study is to compare urine iodine levels of participants with/without periodontitis.

The main question it aims to answer is there a relationship between iodine levels of urine and periodontitis.

Participants will give urine samples without any intervention.

DETAILED DESCRIPTION:
Periodontitis is a chronic, inflammatory disease with a cyclical course with active and passive periods, which may result in the destruction of gingival fibers, resorption of alveolar bone, and subsequent tooth loss, by spreading the inflammatory event that started in the gingiva to the tissues supporting the tooth as a result of the effects of bacteria. The disease is closely associated with many systemic conditions. These conditions include diabetes, cardiovascular diseases, respiratory diseases, birth complications, pregnancy, puberty.

Iodine deficiency is an important public health problem by affecting 10-15% of the population due to the diseases it causes. Iodine deficiency affects individuals of all ages. When the daily iodine requirement cannot be met, a group of mental, physical and developmental retardation symptoms called "Iodine deficiency disorders" (IEB) (Iodine deficiency disorders-IDD) occur. With the obligatory iodization of table salt, which started in 1998 in order to eliminate iodine deficiency in Turkey, this problem has been tried to be combated by switching to iodized salt consumption.

The study material was used by 73 adult individuals who applied to Atatürk University Faculty of Dentistry, Department of Periodontology for different reasons {1. group (H): periodontally healthy individuals, group 2 (P): individuals with periodontitis}. Urine samples will be collected from the participants without any periodontal intervention. Iodine levels in the urine will be studied.

There are studies in the literature to determine iodine deficiency and to determine the population periodontal disease status; however, there are no studies evaluating the possible relationship between iodine deficiency and periodontitis.

The aim of this study; To evaluate the iodine levels detected in the urine samples of patients with periodontitis by comparing them with healthy controls, and to investigate the possible role of iodine deficiency in the pathogenesis of periodontitis or a simple marker of disease activity in the light of these findings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals should not have any systemic disease that may or may not require medication, including salivary gland pathologies, and not particularly thyroid organ pathologies.
* Individuals have not been continuously treated with anti-inflammatory, antioxidant or similar drugs in the last 6 months,
* Individuals have not received periodontal treatment until 6 months ago,
* Individuals must have at least 14 teeth
* Patients diagnosed with stage 3 periodontitis

Exclusion Criteria:

* Having a systemic disease such as cardiovascular, diabetes, hypertension, thyroid organ pathologies, chronic kidney failure
* Being pregnant/breastfeeding
* Being on medication for any reason
* Being a smoker/tobacco user
* Having another periodontal disease other than periodontitis
* Having a chronic inflammatory disease (COPD, asthma)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals who referred to Atatürk University, Department of Periodontology
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
iodine deficiency | 0-1 hours of the diagnosis
  iodine level of participants

CONTACTS AND LOCATIONS:
Overall Officials: DİDEM ÖZKAL EMİNOĞLU, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided